CLINICAL TRIAL: NCT01424020
Title: Estimation de la capacité Fonctionnelle à la Marche Par Questionnaire Clinique Chez Les Patients adressés Pour Bilan artériel Des Membres inférieurs
Brief Title: Walking Estimated Limitation Calculated by History - Study 2
Acronym: WELCH-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-P 2011-06
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Peripheral Artery Disease
Keywords: Questionnaire; peripheral artery disease; execise
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- questionnaire (Experimental): Patients suspected of peripheral artery disease and, as such, referred for a vascular investigations and submitted the WELCH questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Self completed questionnaire, Supervised by the physician Ankle brachial index (ABI) calculation Maximal walking distance (MWD) on treadmill or over the 6 minutes walking test (when available)
  Other Names: Walking impairment questionnaire (WIQ); Walking estimated limitation calculated by history (WELCH)

SUMMARY:
The purpose of this study is to test and validate a new questionnaire in order to get a "walking estimated limitation calculated by history (WELCH) in patients referred for vascular investigations.

DETAILED DESCRIPTION:
Two questionnaires the WELCH and the "walking impairment questionnaire" (WIQ) are submitted to patients referred for vascular investigations for suspêcted peripheral arterial disease (PAD). Comparison of score to hemodynamic parameters (first goal) or maximal walking distance (MWD) on treadmill (secondary goal). Scoring of the WIQ is performed according to references. Scoring of the WELCH has been submitted for copyright protection (involves a series of 4 additions a subtraction and a single multiplication)

ELIGIBILITY:
Inclusion Criteria:

* French Native language
* 18 years old or older
* Signed consent
* Covered by the French social care system

Exclusion Criteria:

* Unable to participate for administrative reasons
* Psychiatric troubles
* Pain at rest or critical limb ischemia
* Unable to walk (ex: wheelchair subjects)

Note: previous inclusion in the protocole is note an exclusion criterion for a new participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2011-09; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of questionnaires with errors after self completion | 1 day
  Analysis of first inclusion only in patients that are included multiple times over the study period. Predetermined score for the WELCH questionnaire answers [(4 items); (4 additions & 1 multiplication)] and WIQ... estimation of the percentage of errors with 95% confidence interval. Comparison of the two percentages

SECONDARY OUTCOMES:
Correlation with ankle brachial index (ABI) | 1 day
  Analysis of first inclusion only in patients that are included multiple times over the study period. Calculation of questionnaire scores from predetermined methods and analysis of the coefficient of determination and coefficient of correlation to minimal ABI
Correlation with treadmill result | 1 day
  Analysis of first inclusion only in patients that are included multiple times over the study period.Calculation of questionnaires score from predetermined methods and analysis of the coefficient of determination and coefficient of correlation to maximal walking distance on treadmill, in the subgroup of patients that have a routine treadmill scheduled during the visit.
Facility of the scoring of the questionnaires | 1 day
  Proportion of WELCH scores calculated by physician and comparison to the proportion of WIQ score calculated by physicians as a estimation of the facility to calculate the score by mental calculation in routine
Reliability of the questionnaire | 3 weeks
  Comparison of the scores of the WELCH in the patients that may be seens within 3 weeks of their first inclusion, for any reasons, (e.i. seen first for a doppler and two weeks later for a treadmill test)over the study period. Analysis of the reliability through the coefficient of variation of the score.
sensitivity of the WELCH to changes | 1 year
  Comparison of the scores of the WELCH in the patients that may be seens within 1 year from their first inclusion, for any reasons, (e.i. seen follow up of their disease)over the study period. Analysis of the changes of the score to changes of the ABI. Analysis of the changes of the score to changes in maximal walking distance if available.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — University Hospital in Angers
Locations (18):
- France (18):
  - Vascular investigation, Angers
  - Vascular Medicine, Annecy
  - Vascular Medicine, Aubenas
  - Rehabilitation, Ballan-Miré
  - Vascular Medicine, Belfort
  - Vascular Medicine, Caen
  - Vascular Medicine, Castanet-Tolosan
  - Vascular Medicine, Champagnole
  - Vascular Medicine, Chazelles-sur-Lyon
  - Rehabilitation, Hauteville
  - Vascular Medicine, Paris
  - Vascular Medicine, Perpignan
  - Vascular Medicine, Périgueux
  - Vascular Medicine, Reims
  - Vascular Medicine, Sallanches
  - Vascular Medicine, Tarbes
  - Vascular Medicine, Villenave-d'Ornon
  - Vascular Medicine, Wattrelos